CLINICAL TRIAL: NCT03937115
Title: Effets de la tDCS Sur la Performance Sportive de 2 Profils d'athlètes : Explosifs (Sauteurs de Haut Niveau et Amateur) et Endurants (Cyclistes de Haut Niveau et Amateur)
Brief Title: Effect of tDCS on Sport Performance for Two Categories of Athletes : Explosive Profile and Enduring Profile
Acronym: COMPETE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: API/2018/97
Record Dates: First submitted 2019-03-06; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers; High-level Sportsman
Keywords: tDCS; Noninvasive brain stimulation; Endurance performance; Cognitive performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group S1 (Experimental): High level jump practice : more 4000 hours of practice during the last five years
  Interventions: Device: Active tDCS; Device: Sham tDCS
- Group S2 (Experimental): Amateur jump practice : less 4000 hours of practice during the last five years
  Interventions: Device: Active tDCS; Device: Sham tDCS
- Group C1 (Experimental): High level cycling practice: more 4000 hours of practice during the last five years
  Interventions: Device: Active tDCS; Device: Sham tDCS
- Group C2 (Experimental): Amateur cycling practice: less 4000 hours of practice during the last five years
  Interventions: Device: Active tDCS; Device: Sham tDCS
- Group T (Experimental): Sedentary : less two hours of recreationally practice of sport by week
  Interventions: Device: Active tDCS; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — 2 active tDCS sessions (20 min each, 2 mA) applied to the dlPFC and right motor cortex
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: Group S1; Group S2
Device: Sham tDCS — 1 sham tDCS session (20 min, 0 mA) applied to the dlPFC
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: Group S1; Group S2
Device: Active tDCS — 10 tDCS sessions (2 sessions/day for 5 days, 20 mA, 20 min each) applied to the dlPFC
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: Group C1; Group C2; Group T
Device: Sham tDCS — 10 tDCS sessions (2 sessions/day for 5 days, 0 mA, 20 min each) applied to the dlPFC
  Other Names: Starstim® (Neuroelectrics, Spain)
  Arms: Group C1; Group C2; Group T

SUMMARY:
The study aims to compare the effects of tDCS applied on the dorsolateral prefrontal cortex (dlPFC) vs sham on the neuromuscular system. Two types of athletes will benefit from stimulation: jumper and cyclists. Short and long term effects are assesed by electromyographic records, experimental tasks and self-rated scales.

DETAILED DESCRIPTION:
Transcranial direct current stimulation is a technique of noninvasive brain stimulation which delivers a electrical current to the scalp to modulate the neuronal activity. Depending on the polarity of stimulation, tDCS induces a neural hyperexcitability (with anode) or hypoexcitability (with cathode) of the target area.

Due to its neuromodulatory action, ease of use and low safety, tDCS can be used as a potential treatment but also as an investigative tool in neurophysiology. Thus, studies have shown a beneficial effect of tDCS on cognitive and motor functions. Nevertheless, studies conducted on motor performance and the reduction of neuromuscular fatigue show disparate results. It is impossible to conclude whether tDCS allows for improved performance and is a means of doping.

With a prospective, sham-controlled, crossover, double-blind design, this study aims to evaluate the effect of tDCS on neuromuscular fatigue resistance during explosive (jumping) and endurance (cycling) exertion.

This study is divided into two parts:

* Part A: jumping group
* Part B: cycling group.

During Part A, participants visit the laboratory on 3 occasions. Each visit is organized in the same way and is at least 48 hours apart from the previous one.

Participants are divided into two groups according to their level of experience (amateurs vs. high level).

Before the session of tDCS, participants carry out a psychometric assessment (MCQ, BIS10) and experimental tasks (BART, EEFRT, STROOP test and Go NoGo task). Then, they performed three types of jumps (long jump, squat jump and countermovement jump). Finally, participants benefit from neuromuscular tests (EMG recording of plantar flexor muscle activity, percutaneous stimulation of the posterior tibial nerve).

Subjects will be submitted to three sessions of tDCS (2 actives and one sham), one by visit, in the order of randomization. Current intensity will be of 2 mA (or 0 mA), through 25 cm² surface electrodes, during 20 minutes. The positioning of the stimulation electrodes will be carried out in compliance with EEG 10/20 standards:

- Sequence order determined by randomization:

1. Anode: F3 / Cathode: AF8/ Stimulation intensity: 2 mA
2. Anode: F3/ Cathode: AF8/ Stimulation intensity: 0 mA
3. Anode: FC2/ Cathode: Left shoulder/ Stimulation intensity: 2 mA

Immediately after the stimulation, participants perform motor and cognitive task again and the results are compared.

During part B, subjects participate in two training sessions of five days each. The training sessions are one month apart.

Participants are divided into three groups according to their level of experience (amateurs vs. high level vs. sedentary).

Each day, the subjects perform two twenty-minute time trials during which they receive a session of tDCS. (one week with the active tDCS, one week with the sham). So, subjects will be submitted to 10 tDCS stimulation sessions (active or sham) for five consecutive days (2 sessions of 20 minutes/day). Current intensity will be of 2 mA, through 25 cm² surface electrodes, placed over the dlPFC and the supraorbital region (anode position over F3 and cathode over AF8, according to the EEG 10-20 international system).

At J1 and J5 of each session (before and after session training), subjects carry out a psychometric assessment (MCQ, BIS10) and experimental tasks (BART, EEFRT, STROOP test and Go NoGo task) and benefit from neuromusculars tests (EMG recording of plantar flexor muscle activity, percutaneous stimulation of the posterior tibial nerve). Baseline measures will be compared to those obtained immediately after the end of sessions (5 days: short-term effects), and to 12 and 30 days later (long-term effects). Active and sham stimulation sessions outcomes will as well be compared.

ELIGIBILITY:
Inclusion Criteria:

* Man older than 18 years old
* Right-handed
* Signed informed Consent form
* Subject affiliated to or beneficing from a French social security regime
* According to groups :

  * Part A :

    * Group S1 : High level jump practice : more 4000 hours of practice during the last five years
    * Group S2 : Amateur jump practice : less 4000 hours of practice during the last five years
  * Part B :

    * Group C1 : High level cycling practice: more 4000 hours of practice during the last five years
    * Group C2 : Amateur cycling practice: less 4000 hours of practice during the last five years
    * Group T : Sedentary : less two hours of recreationally practice of sport by week

Exclusion Criteria:

* Younger than18 years old
* Left-handed
* Subject under measure of protection or guardianship of justice
* Subject beneficiary from a legal protection regime
* Subject unlikely to cooperate or low cooperation stated by investigator
* Subject not covered by social security
* Suject with comorbidities : addictive (except : tea, coffee, tobacco), psychiatric, severe somatic pathologies (specially tumors, degenerative disease) or progressive neurologic pathologie
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File"

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Performance (in meters) measured during jumps | Day 5
  Performance measurement (in meters) during the three types of jumps (long jump, squat jump and countermovement jump) before and after tDCS session

SECONDARY OUTCOMES:
Average power during the time trial before and after 10 tDCS sessions | Day 35
  Average power (in watts) measured during a 20min time trial before and after 10 tDCS sessions for 5 days
BIS-10 scores | Day 60
  Compared scores from the French version of the Barratt Impulsiveness Scale (BIS-10). The French version of the BIS-10 is a self-rated 34 item questionnaire, composed by three subscales: motor-impulsivity, cognitive-impulsivity and non-planning-impulsivity. Each item is scored on a 0 to 4 points scale. Higher scores indicate higher levels of impulsivity.
MCQ scores | Day 60
  Compared scores from the French version of the Monetary Choice Questionnaire. The MCQ is a self-rated 27 item questionnaire which assessed the discounting. Delay discounting is the decline in the present value of a reward with delay to its receipt.
  Example item: " Would you prefer 25€ today or 75€ in 15 days? "
  For each item, subjects must choose between a low immediate reward and a higher delayed reward.
  Waiting times vary from 7 days to 186 days, and rewards are divides into 3 magnitudes: low (25-35€), medium (50-60€), high (75-85€).
  This will allow assessing:
  * the influence of the the magnitude of the difference between the two rewards proposed,
  * the impact of the time on the reward's subjective value (speed at which the reward is devalued over time), reflected in the k index.
  This index is calculated separately for each magnitude, and an average index is calculated for each subject.
  The more the k index is high, the more the subject is considered impulsive.
Stroop task | Day 60
  Compared results from the experimental Stroop task, assessing response inhibition.
Go/No-Go task | Day 60
  Compared results from the experimental Go/No-Go task, assessing response inhibition.
Effort Expenditure for Reward Task | Day 60
  Compared results from the experimental Effort Expenditure for Reward Task, assessing motivation
Balloon Analog Risk Task | Day 60
  Compared results from the experimental Balloon Analog Risk task, assessing impulsivity
QIDS-C16 scale | Day 60
  Compared scores from the French version of the Quick Inventory of Depressive Symptomatology. The QIDS-C16 is a 16 item questionnaire completed by the clinician to assess the depressive symptomatology and the severity of the depression.
  These 16 items are constructed around the 9 following symptoms:
  * sad mood,
  * concentration,
  * autocriticism,
  * suicidal thoughts,
  * ahnedonia,
  * fatigue,
  * sleep disorders,
  * appetite/weight changes,
  * psychomotor retardation/agitation. This scaled is based on the intensity of each symptom in the 7 last days, regardless of its chronicity or its recent apparition.
  Each symptom is rated 0 to 3. The total score thus vary from 0 to 27.
QIDS-SR16 scale | Day 60
  Compared scores from the French version of the Quick Inventory of Depressive Symptomatology. The QIDS-SR16 is a self-rated 16 item questionnaire, assessing the intensity of depressive symptomatology.
  These 16 items are constructed around the 9 following symptoms:
  * sad mood,
  * concentration,
  * autocriticism,
  * suicidal thoughts,
  * ahnedonia,
  * fatigue,
  * sleep disorders,
  * appetite/weight changes,
  * psychomotor retardation/agitation. This scaled is based on the intensity of each symptom in the 7 last days, regardless of its chronicity or its recent apparition.
  Each symptom is rated 0 to 3. The total score thus vary from 0 to 27.

CONTACTS AND LOCATIONS:
Overall Officials: Djamila BENNABI, MD, Principal Investigator — CHU de Besançon
Locations (2):
- France (2):
  - CHU Besancon - Clinical Psychiatric Department, Besançon
  - EA4660- C3S, Culture, Sport, Santé, Société, Besançon

REFERENCES:
- [Derived] Grandperrin Y, Grospretre S, Nicolier M, Gimenez P, Vidal C, Haffen E, Bennabi D. Effect of transcranial direct current stimulation on sports performance for two profiles of athletes (power and endurance) (COMPETE): a protocol for a randomised, crossover, double blind, controlled exploratory trial. Trials. 2020 Jun 3;21(1):461. doi: 10.1186/s13063-020-04412-0. PMID 32493462